CLINICAL TRIAL: NCT06599463
Title: Efficacy Assessment of Lenvatinib Associated with Pembrolizumab in Metastatic Endometrial Cancer: a French Multicentric Retrospective Early Access Program-based Study
Acronym: LARENA
Status: Completed | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: GINECO-EN204; RECF-005767 (Registry Identifier: INCA)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Endometrial Cancer
Keywords: metastatic; endometrial; cancer; endometrial cancer; metastatic cancer
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
LARENA is a multicentric retrospective study (secondary use of data) of consecutive patients prospectively registered in the lenvatinib plus pembrolizumab French early access program (Temporary Authorisation for Use). The source of data will be the patient's medical file. We will manually review all files of the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients having received at least one dose of lenvatinib plus pembrolizumab in the context of the French early access program (Temporary Authorisation for Use) approved by the French Health Autority.
* Patients with advanced or recurrent endometrial cancer whose disease is progressing during or following prior platinum-based chemotherapy at any stage and who are not eligible for curative surgery or radiotherapy, according to the French early access program (Temporary Authorisation for Use) approved by the French Health Autority criteria.

Exclusion Criteria:

* Patients who refuse the collection and use of their personal data in the course of this research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who received lenvatinib with pembrolizumab in metatstatic endometrial cancer.
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Median progression free survival (PFS) | An estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the first administration of lenvatinib + pembrolizumab to the date of the first documented disease progression according to RECIST1.1 or death due to any cause whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | An estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the initial diagnosis of metastatic endometrial cancer to the date of death
Clinical benefit rate (CBR: SD, CR, PR). | An estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the first administration of lenvatinib + pembrolizumab to the date of the first documented disease progression according to RECIST1.1 or death due to any cause whichever occurs first.
Safety according to NCI CTCAE criteria v5.0. | An estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the first administration of lenvatinib + pembrolizumab to the date of the first documented disease progression according to RECIST1.1 or death due to any cause whichever occurs first.
Frequency and type of oncogeriatric testing. | an estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the first administration of lenvatinib + pembrolizumab to the date of the first documented disease progression according to RECIST1.1 or death due to any cause whichever occurs first.
Objective response rate (ORR: CR, PR) | An estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the first administration of lenvatinib + pembrolizumab to the date of the first documented disease progression according to RECIST1.1 or death due to any cause whichever occurs first.
PFS with lenvatinib+pembrolizumab according to MMR/MSI status. | An estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the first administration of lenvatinib + pembrolizumab to the date of the first documented disease progression according to RECIST1.1 or death due to any cause whichever occurs first.
Frequency and type of medical and paramedical follow-up procedures. | an estimated median follow-up of 5 months from March 2022 to May 2024.
  Time from the first administration of lenvatinib + pembrolizumab to the date of the first documented disease progression according to RECIST1.1 or death due to any cause whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Diana BELLO ROUFAI, Principal Investigator — Institut Curie
Locations (24):
- France (24):
  - ICO Paul Papin, Angers
  - Sainte Catherine - Institut du Cancer Avignon, Avignon
  - CHU Jean Minjoz, Besançon
  - ICONE, Bezannes
  - Clinique TIVOLI, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU de DIJON, Dijon
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Hôpital Européen George Pompidou, Paris
  - Centre CARIO-HPCA, Plérin
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - CHI de Cornouaille, Quimper
  - Centre Eugène Marquis, Rennes
  - Institut Curie, Saint-Cloud
  - CHU Saint-Etienne - Hôpital Bellevue, Saint-Etienne
  - ICANS, Strasbourg
  - Oncopole Claudius Regaud - IUCT Oncopole, Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
  - Centre Hospitalier de Valence, Valence

IPD SHARING:
Plan to Share IPD: No